CLINICAL TRIAL: NCT00001391
Title: Bone Regeneration Using Bone Marrow Stromal Cells
Status: Completed | Type: Observational
Sponsor: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 940188; 94-D-0188
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2010-10-04

CONDITIONS: Bone Disease; Craniofacial Abnormality; Healthy
Keywords: Augmentation; Osteogenesis; Stem Cells; Bone Formation; Bone Induction
MeSH Terms: conditions — Bone Diseases; Craniofacial Abnormalities

SUMMARY:
Deficient or inappropriate healing of bone impacts clinical decision-making and treatment options in orthopedics, oral and maxillofacial surgery, plastic surgery and periodontics. While a number of auto- and allografting techniques have been used to regenerate craniofacial defects caused by infective, neoplastic or trauma-induced bone loss, each method has significant limitations. Our research group in the Craniofacial and Skeletal Diseases Branch of NIDCR has developed methods to culture and expand cell populations derived from mouse bone marrow stroma. We believe that an important next step is to apply the information gained in animal studies to treat osseous defects in humans. We propose to examine the potential of cultured human bone marrow stromal cells to serve as an abundant source of osteoblastic progenitor cells. These cells will ultimately be used to graft craniofacial osseous defects. In the course of this study we will: (1) develop methods for the propagation and enrichment of osteoblastic progenitor cells from bone marrow stroma; (2) test various vehicles for the transfer of bone marrow stromal cells to osseous defects in recipient animals; (3) determine optimal culturing and transplantation conditions for the eventual transplantation of bone marrow stromal cells into human recipients. These studies will define the parameters of bone marrow stromal cell transplantation and will generate models for future therapeutic strategies.

DETAILED DESCRIPTION:
Deficient or inappropriate healing of bone impacts clinical decision-making and treatment options in orthopedics, oral and maxillofacial surgery, plastic surgery and periodontics. While a number of auto- and allografting techniques have been used to regenerate craniofacial defects caused by infective, neoplastic or trauma-induced bone loss, each method has significant limitations. Our research group in the Craniofacial and Skeletal Diseases Branch of NIDCR has developed methods to culture and expand cell populations derived from mouse bone marrow stroma. We believe that an important next step is to apply the information gained in animal studies to treat osseous defects in humans. We propose to examine the potential of cultured human bone marrow stromal cells to serve as an abundant source of osteoblastic progenitor cells. These cells will ultimately be used to graft craniofacial osseous defects. In the course of this study we will: (1) develop methods for the propagation and enrichment of osteoblastic progenitor cells from bone marrow stroma; (2) test various vehicles for the transfer of bone marrow stromal cells to osseous defects in recipient animals; (3) determine optimal culturing and transplantation conditions for the eventual transplantation of bone marrow stromal cells into human recipients. These studies will define the parameters of bone marrow stromal cell transplantation and will generate models for future therapeutic strategies.

ELIGIBILITY:
* INCLUSION CRITERIA:

Males and females 18 years and older.

EXCLUSION CRITERIA:

Subjects may not have metabolic bone diseases, pregnancy or taking drugs affecting skeletal metabolism.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 1994-08-03; Study Completion 2010-10-04

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Owen M, Friedenstein AJ. Stromal stem cells: marrow-derived osteogenic precursors. Ciba Found Symp. 1988;136:42-60. doi: 10.1002/9780470513637.ch4. PMID 3068016
- [Background] Krebsbach PH, Kuznetsov SA, Satomura K, Emmons RV, Rowe DW, Robey PG. Bone formation in vivo: comparison of osteogenesis by transplanted mouse and human marrow stromal fibroblasts. Transplantation. 1997 Apr 27;63(8):1059-69. doi: 10.1097/00007890-199704270-00003. PMID 9133465
- [Background] Dahlin C, Linde A, Gottlow J, Nyman S. Healing of bone defects by guided tissue regeneration. Plast Reconstr Surg. 1988 May;81(5):672-6. doi: 10.1097/00006534-198805000-00004. PMID 3362985